CLINICAL TRIAL: NCT05192161
Title: Computational Medical Imaging (Radiomics) and Prediction of Diffusion/FLAIR Mismatch in Stroke Patients
Brief Title: Computational Medical Imaging and Prediction of Diffusion/FLAIR Mismatch in Stroke Patients
Acronym: RADIOMIXSTROKE
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: RADIOMIXSTROKE
Record Dates: First submitted 2021-12-30; First posted 2022-01-14 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Stroke is a public health issue and a priority for our institution. MRI plays an essential role in the management of stroke. In this context, the contribution of MRI is diagnostic, etiological and prognostic.

Among the MRI parameters evaluated in the acute phase of the stroke, the evaluation of the mismatch between the DIFFUSION and FLAIR sequences is crucial as it will directly contribute to the therapeutic decision. A FLAIR-diffusion mismatch, i.e., a lesion with a diffusion but not a FLAIR hypersignal, identifies patients whose time of onset of symptoms is probably less than 4.5 hours. It is therefore understandable that the main arterial recanalization techniques performed in the acute phase are primarily reserved for patients with a positive mismatch.

In current practice, mismatch assessment is performed subjectively, by visually comparing the two sequences, which is known to be the cause of a lack of reproducibility and diagnostic performance.

Computational medical imaging techniques ("radiomics") have recently gained momentum and offer the prospect of automated and therefore more reproducible analysis of medical imaging data. In stroke patients, radiomics extracted from FLAIR imaging could thus contribute to describe the "diffusion flair" mismatch in a continuous and objective way.

For the time being, data analysis cannot be performed in real time due to technical constraints. If it is proven that radiomics can reliably analyze the mismatch on the FLAIR sequence alone, the next step will be to make the analysis feasible in clinical routine (i.e. in a time frame adapted to the therapeutic management).

ELIGIBILITY:
Inclusion Criteria:

* Patient with age ≥ 18 years
* Patient with supra-tentorial stroke treated by mechanical thrombectomy and who had MRI imaging on admission before endovascular treatment at Paris Saint-Joseph Hospital
* Complete MRI protocol including Diffusion and FLAIR sequences
* French-speaking patient

Exclusion Criteria:

* Patient under guardianship or curatorship
* Patient deprived of liberty
* Patient under court protection
* Patient objecting to the use of his data for this research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred for suspected stroke between January 1, 2016 and May 1, 2021 at Paris Saint Joseph Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2023-04-05 (Actual); Primary Completion 2023-05-05 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
ability of a computational medical imaging technique ("radiomics"), performed on the FLAIR sequence alone, to predict the FLAIR diffusion mismatch in patients with ischemic stroke | Day 1
  This outcome corresponds to FLAIR / Diffusion mismatch scores estimated with both techniques: automated and visual analysis.

SECONDARY OUTCOMES:
Inter-technique comparison of mismatch assessment between automated "radiomics" analysis and subjective visual analysis (currently performed in clinical routine) | Day 1
  This outcome corresponds to the reproducibility and inter-technical agreement on the extent of the mismatch.
Evaluation of the prognostic value of the scores obtained with the two methods | Month 3
  This outcome corresponds to the correlation of the scores obtained with the Rankin score at 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Jerome HODEL, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (2):
- France (2):
  - CHRU Lille, Lille
  - Groupe Hospitalier Paris Saint-Joseph, Paris

REFERENCES:
- [Background] Powers WJ, Rabinstein AA, Ackerson T, Adeoye OM, Bambakidis NC, Becker K, Biller J, Brown M, Demaerschalk BM, Hoh B, Jauch EC, Kidwell CS, Leslie-Mazwi TM, Ovbiagele B, Scott PA, Sheth KN, Southerland AM, Summers DV, Tirschwell DL; American Heart Association Stroke Council. 2018 Guidelines for the Early Management of Patients With Acute Ischemic Stroke: A Guideline for Healthcare Professionals From the American Heart Association/American Stroke Association. Stroke. 2018 Mar;49(3):e46-e110. doi: 10.1161/STR.0000000000000158. Epub 2018 Jan 24. PMID 29367334
- [Background] Thomalla G, Cheng B, Ebinger M, Hao Q, Tourdias T, Wu O, Kim JS, Breuer L, Singer OC, Warach S, Christensen S, Treszl A, Forkert ND, Galinovic I, Rosenkranz M, Engelhorn T, Kohrmann M, Endres M, Kang DW, Dousset V, Sorensen AG, Liebeskind DS, Fiebach JB, Fiehler J, Gerloff C; STIR and VISTA Imaging Investigators. DWI-FLAIR mismatch for the identification of patients with acute ischaemic stroke within 4.5 h of symptom onset (PRE-FLAIR): a multicentre observational study. Lancet Neurol. 2011 Nov;10(11):978-86. doi: 10.1016/S1474-4422(11)70192-2. Epub 2011 Oct 4. PMID 21978972
- [Background] Qiu W, Kuang H, Nair J, Assis Z, Najm M, McDougall C, McDougall B, Chung K, Wilson AT, Goyal M, Hill MD, Demchuk AM, Menon BK. Radiomics-Based Intracranial Thrombus Features on CT and CTA Predict Recanalization with Intravenous Alteplase in Patients with Acute Ischemic Stroke. AJNR Am J Neuroradiol. 2019 Jan;40(1):39-44. doi: 10.3174/ajnr.A5918. Epub 2018 Dec 20. PMID 30573458
- [Background] Chen Q, Xia T, Zhang M, Xia N, Liu J, Yang Y. Radiomics in Stroke Neuroimaging: Techniques, Applications, and Challenges. Aging Dis. 2021 Feb 1;12(1):143-154. doi: 10.14336/AD.2020.0421. eCollection 2021 Feb. PMID 33532134
- [Background] Tang TY, Jiao Y, Cui Y, Zhao DL, Zhang Y, Wang Z, Meng XP, Yin XD, Yang YJ, Teng GJ, Ju SH. Penumbra-based radiomics signature as prognostic biomarkers for thrombolysis of acute ischemic stroke patients: a multicenter cohort study. J Neurol. 2020 May;267(5):1454-1463. doi: 10.1007/s00415-020-09713-7. Epub 2020 Feb 1. PMID 32008072
- [Background] Feng R, Badgeley M, Mocco J, Oermann EK. Deep learning guided stroke management: a review of clinical applications. J Neurointerv Surg. 2018 Apr;10(4):358-362. doi: 10.1136/neurintsurg-2017-013355. Epub 2017 Sep 27. PMID 28954825